CLINICAL TRIAL: NCT00930124
Title: Distraction Versus Orthognathic Surgery - Which One is Better for Cleft Palate Patients
Brief Title: Cleft Orthognathic Surgery Versus Distraction Osteogenesis - Which is Better?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Lim K Cheung, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP_DOvsCO
Record Dates: First submitted 2009-01-21; First posted 2009-06-30 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Cleft Lip and Palate; Maxillary Hypoplasia
Keywords: cleft lip and palate; distraction osteogenesis; conventional orthognathic surgery; stability; morbidity; soft tissue changes; psychological adjustment; speech changes; velopharyngeal function
MeSH Terms: conditions — Cleft Lip; Retrognathia | interventions — Orthognathic Surgery; Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group 1 will receive Conventional orthognathic surgery
  Interventions: Procedure: Orthognathic surgery
- 2 (Active Comparator): Group 2 will receive distraction osteogenesis
  Interventions: Procedure: Distraction osteogenesis

INTERVENTIONS:
Procedure: Orthognathic surgery — Patients with moderate maxillary hypoplasia needing an advancement of 4-10mm
  Other Names: cleft osteotomy
  Arms: 1
Procedure: Distraction osteogenesis
  Other Names: cleft distraction
  Arms: 2

SUMMARY:
Cleft lip and palate patients normally present with a sunken face due to collapse in the middle part of the face and inability of the upper and lower teeth to meet during chewing. This situation constitutes a serious aesthetic and mastication problem. A single surgical operation known as orthognathic surgery was traditionally performed to move the upper jaw forward to a more normal position and allow chewing function to be regained. However, due to scar tissue from the original surgical repair of the cleft palate, this procedure is known to be unstable causing bone to rapidly go back to its original position. A new concept of moving the upper jaw bone gradually by 1mm per day using a special device attached to the bone called distraction osteogenesis was established in 1996. Animal studies have shown that this technique can produce stable results with minimal relapse. The feasibility of correcting cleft deformities by gradual distraction has been confirmed by our own clinical studies. The aim of this study (which is the first of its kind) is to conduct a prospective randomized controlled study and compare the treatment outcomes of the current standard (orthognathic surgery) with distraction osteogenesis (gradual bone movement). The objectives focus on four aspects: morbidity, stability, speech function and psychological impact. The results from this study will clarify several clinical dilemmas in decision making when choosing whether to use orthognathic surgery or distraction osteogenesis in the treatment of cleft lip and palate patients. In addition, it will also inform our multidisciplinary research team to improve the total care of the cleft lip and palate patients.

Gradual bone distraction of the midface in cleft palate patients is more stable, less detrimental to speech, and no more troublesome to the patient than conventional osteotomy and bone transposition (orthognathic surgery).

DETAILED DESCRIPTION:
Maxillary hypoplasia leading to sunken midface is a common developmental problem in CLP patients and is related to a combination of congenital reduction in midfacial growth and the surgical scar from the repair of the cleft palate. Therefore CLP patients commonly present with short midface and narrow hard palate and severe malocclusion.

Conventional orthognathic surgery can advance, expand and lengthen the maxilla to a normal position in relation to the skull and the occlusion. However, such immediate surgical transposition of the cleft maxilla is technically difficult due to the severe deformity demanding large surgical movement and the tension from the palatal scar. Studies have demonstrated that the repositioned maxilla is rather unstable in the long term. In addition, velopharyngeal competence could be compromised by this immediate advancement technique resulting in abnormally nasal speech.

The feasibility of gradual lengthening of the under-developed mandible in syndromal patients by distraction osteogenesis has been proven. The gradual movement of the maxilla activated by the implanted distractors can theoretically overcome the tension from the palatal scar and the soft palate musculature. This may reduce the long term skeletal relapse of the cleft maxilla and the speech distortion. On the other hand, the distraction procedures involve the surgical insertion and removal operations and the retention of the devices over a two month period. This may increase the chance of infection, social inconvenience and ultimately affect the patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Cleft lip and palate patients who required maxillary advancement ranging from 4-10 mm

Exclusion Criteria:

* syndromic cases, skeletal maturity not yet reached

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-06; Primary Completion 2004-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
standardized questionnaires, lateral cephalographs,nasoendoscopy, nasometry | intra-operative and post-operatively at 2-6 weeks, 2,3,6,months, 1, 2, 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lim K Cheung, BDS, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- OMFS, Faculty of Dentistry, The University of Hong Kong, Sai Ying Pun, Hong Kong